CLINICAL TRIAL: NCT02330757
Title: Hormone Replacement Therapy Versus Minimal Ovarian Stimulation for Endometrial Preparation Prior to Frozen-thawed Embryo Transfer in Non Polycystic Ovarian Syndrome Patients
Brief Title: HRT Versus MOS for Endometrial Preparation Prior to FET in Non PCOS Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSA2
Record Dates: First submitted 2015-01-01; First posted 2015-01-05 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Infertility
Keywords: Frozen-thawed embryo transfer; FET protocols
MeSH Terms: conditions — Infertility | interventions — Estradiol; Gonadotropins; Menotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HRT group (Active Comparator): Women will be subjected to HRT using Estradiol valerate before FET
  Interventions: Drug: Estradiol valerate
- MOS group (Active Comparator): Women will be subjected to MOS using sequential clomiphene citrate and gonadotropin before FET
  Interventions: Drug: Sequential Clomiphene citrate and Gonadotropin

INTERVENTIONS:
Drug: Estradiol valerate — Women will be given estradiol valerate 4 mg daily from day 2 to day 12 of the cycle then the endometrial thickness will be assessed on day 13 by transvaginal sonography (TVS). If the endometrium is ≥ 8 mm and of moderate echogenicity, luteal phase support (using progesterone supplements) will be started but if the endometrium is < 8 mm, estradiol valerate will be continued until reaching appropriate endometrial thickness and echogenicity then the luteal phase support will be started.
  Other Names: Cycloprogynova (white tablets)
  Arms: HRT group
Drug: Sequential Clomiphene citrate and Gonadotropin — Women will be given clomiphene citrate in dose of 100-150 mg daily for 5 days (from day 2 to day 6 of the cycle) then switched to low dose gonadotropin (75-150 IU daily) followed by monitoring of the follicular growth (folliculometry) ); starting from day 10 of the stimulation cycle and repeated every 2 days. Final oocyte maturation will be induced by administration of human chorionic gonadotropin (HCG) when there will be at least one leading follicle > 18 mm in diameter followed by luteal phase support (using progesterone supplements) after 48 hours.
  Other Names: Sequential Clomid and Menogon
  Arms: MOS group

SUMMARY:
Evaluation of endometrial preparation using either hormonal therapy or ovarian stimulation prior to frozen-thawed embryo transfer (FET) in patients without polycystic ovarian syndrome (PCOS)

DETAILED DESCRIPTION:
Women will be randomly divided into two groups; one will be subjected to endometrial preparation by hormone replacement therapy (HRT) and the other will be subjected to minimal ovarian stimulation (MOS). Women in the HRT group will be given estradiol valerate 4 mg daily from day 2 to day 12 of the cycle then the endometrial thickness will be assessed on day 13 by transvaginal sonography (TVS). If the endometrium is ≥ 8 mm and of moderate echogenicity, luteal phase support (using progesterone supplements) will be started but if the endometrium is < 8 mm, estradiol valerate will be continued until reaching appropriate endometrial thickness and echogenicity then the luteal phase support will be started. Women in the MOS group will be given clomiphene citrate in dose of 100-150 mg daily for 5 days (from day 2 to day 6 of the cycle) then switched to low dose gonadotropin (75-150 IU daily) followed by monitoring of the follicular growth (folliculometry) ); starting from day 10 of the stimulation cycle and repeated every 2 days. Final oocyte maturation will be induced by administration of human chorionic gonadotropin (HCG) when there will be at least one leading follicle > 18 mm in diameter followed by luteal phase support (using progesterone supplements) after 48 hours. In both groups, FET will be planned in the appropriate day according to the stage that the embryos have been cryopreserved in it.

ELIGIBILITY:
Inclusion Criteria:

* Women without PCOS as defined by the Rotterdam criteria.
* Presence of at least 2 cryopreserved good quality cleavage-stage embryo (good quality cleavage-stage embryos display stage-specific cell division, have blastomeres of fairly equal size with few to no cytoplasmic fragments).

Exclusion Criteria:

* PCOS or polycystic ovary on ultrasound scan.
* Moderate or severe endometriosis.
* Hydrosalpinx.
* Uterine abnormalities or myoma.
* Previous uterine surgery.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-10-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 weeks after embryo transfer
  Number of clinical pregnancies (defined as presence of at least one intrauterine gestational sac with fetal pole and cardiac activity on TVS scan at 4-6 weeks after the ET) divided by the number of ET procedures

SECONDARY OUTCOMES:
Implantation rate | 6 weeks after embryo transfer
  Number of gestational sacs on TVS scan at 4-6 weeks after ET divided by the number of transferred embryos
Miscarriage rate | 12 weeks gestational age
  Number of first trimester miscarriages (before 12 weeks gestational age) divided by the number of clinical pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Abdelhafez, Dr, Principal Investigator — Mansoura University
Locations (2):
- Egypt (2):
  - Fertility Care Unit (FCU) in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private fertility care centers, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: Undecided